CLINICAL TRIAL: NCT02970552
Title: A Pilot Study of Vaginal Progesterone to Reduce Preterm Birth Among Women Receiving Antiretroviral Therapy in Pregnancy
Brief Title: Feasibility of Vaginal Progesterone to Reduce HIV-Associated Preterm Birth
Acronym: VP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 16-2174; 1R21HD090987-01 (NIH); Z 31606 (Other: IGHID)
Record Dates: First submitted 2016-11-17; First posted 2016-11-22 (Estimated); Results first posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2019-03

CONDITIONS: PreTerm Birth
Keywords: PreTerm Birth; HIV; Vaginal Progesterone; ART; Adherence; Feasibility
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Vaginal Progesterone (Active Comparator): Daily self-administered vaginal progesterone
  Interventions: Drug: Vaginal Progesterone
- Placebo (Placebo Comparator): Daily self-administered indistinguishable placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vaginal Progesterone — 200 mg micronized vaginal progesterone suppository
  Arms: Vaginal Progesterone
Drug: Placebo — Indistinguishable placebo vaginal suppository
  Arms: Placebo

SUMMARY:
More than 1.5 million HIV-infected women become pregnant each year. Approximately half have access to antiretroviral therapy (ART), but all are at increased risk of preterm birth (PTB). Vaginal progesterone (VP) is a promising and cost-effective intervention to prevent PTB that should be studied in this high-risk population. This pilot study will provide critical insight into the feasibility of a phase III trial by determining whether women are willing to participate, to adhere to study drug, and to complete follow-up.

DETAILED DESCRIPTION:
This will be a mixed method study to evaluate the feasibility and acceptability of a trial of VP to prevent PTB among HIV-infected Zambian women. To assess the feasibility of a full-scale clinical trial, the investigators will implement a pilot two-arm, double-masked, placebo-controlled trial of VP among HIV-infected women in antenatal care in Lusaka, Zambia. Participants will be randomly assigned to either daily self-administered VP or indistinguishable placebo prior to 24 weeks gestational age. In this pilot study, the investigators will be able to estimate study uptake, adherence to study product and protocol, and study retention. To assess the acceptability of a trial to test VP among HIV-infected women in Zambia, the investigators will employ a qualitative approach of longitudinal semi-structured interviews among women agreeing to trial participation and one-time semi-structured interviews (SSIs) among those who decline to participate.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. viable intrauterine pregnancy confirmed by ultrasound
3. presentation to antenatal care prior to 24 weeks gestation
4. antibody-confirmed HIV-1 infection
5. initiating or continuing ART treatment in pregnancy
6. ability and willingness to provide written informed consent
7. willing to adhere to study visit schedule

Exclusion Criteria:

1. multiple gestation
2. non-research indication for antenatal progesterone (i.e. prior spontaneous PTB and/or cervical length <20mm on screening ultrasound)
3. planned or in situ cervical cerclage
4. evidence of threatened abortion, preterm labor, or ruptured membranes
5. major fetal anomaly detected on screening ultrasound
6. known uterine anomaly
7. known or suspected allergy or contraindication to VP or placebo components

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-11-13 (Actual); Study Completion 2018-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Stringer, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Kamwala District Health Centre, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Price JT, Mollan KR, Fuseini NM, Freeman BL, Mulenga HB, Corbett AH, Vwalika B, Stringer JSA. Vaginal progesterone to reduce preterm birth among HIV-infected pregnant women in Zambia: a feasibility study protocol. Pilot Feasibility Stud. 2017 Jul 18;4:21. doi: 10.1186/s40814-017-0170-7. eCollection 2018. PMID 28729911

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vaginal Progesterone | Placebo
Started | 70 | 70
Completed | 67 | 67
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaginal Progesterone | Placebo | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 70 | 70 | 140
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 70 | 140
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 70 | 70 | 140
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Zambia | 70 | 70 | 140

OUTCOME MEASURES:

1. Primary Outcome: Adequate Adherence to Study Product
Description: Number of participants who achieved adequate adherence to study product, defined as proper self-administration of at least 80% of prescribed study product doses, as measured by a dye stain assay of returned applicators
Time Frame: Enrollment through 36th gestational week, an overall total of up to 17 weeks
Population: Participants who returned for at least one follow-up study visit following enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Vaginal Progesterone | Placebo
Number analyzed (Participants) | 68 | 69
Participants | 62 | 63

2. Secondary Outcome: Acceptability of Use of Vaginal Progesterone (VP)
Description: Semi-structured interviews will be held with a random sample of participants who enroll and those who decline enrollment.
Time Frame: At enrollment (20-24 weeks gestation), at 28 weeks gestation, and at 36 weeks gestation
Population: Activation was delayed by 6 months because of a protracted regulatory process. Resulting low resources limited investigators' ability to conduct interviews at all specified times or with decliners. Investigators did conduct a single interview with a sample of participants late in pregnancy or postpartum; these data are captured in outcomes #3 and 4
Arm/Group | Vaginal Progesterone | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Reported Barriers and Facilitators to Adherence to Study Product, Returning Used Applicators, and Retention in the Study
Description: Number of participants reporting barriers and facilitators to study product adherence, returning used applicators, and retention in the study during a semi-structured interview. Participants were selected for an interview based on their overall adherence rates, including those with excellent adherence throughout the study and those with lower adherence rates early or late in their participation. A trained female staff member conducted each 30-minute interview using an interview guide. Interviews were audiotaped, transcribed, and translated into English as necessary.
Time Frame: Late in pregnancy or postpartum
Population: A sample of enrolled participants selected to participate in a semi-structured interview. Investigators included 30 trial participants based on expectations regarding saturation of qualitative themes.
Measure: Count of Participants; unit: Participants
Groups:
- Vaginal Progesterone: Daily self-administered vaginal progesterone Vaginal Progesterone: 200 mg micronized vaginal progesterone suppository
- Placebo: Daily self-administered indistinguishable placebo Placebo: Indistinguishable placebo vaginal suppository
Arm/Group | Vaginal Progesterone | Placebo
Number analyzed (Participants) | 19 | 11
Participants
  Reported any barriers to medication use | 7 | 1
  Discontinued med due to challenges or discomfort | 0 | 0
  Reported any facilitators to medication use | 19 | 11
  Reported barrier to returning used applicators | 0 | 0
  Reported barriers to returning for study visits | 2 | 0
  Reported positive experience with study clinic | 19 | 11

4. Secondary Outcome: Summary of Reported Knowledge, Attitudes, and Practices Related to HIV, Antiretroviral Therapy (ART), Risk of Preterm Birth, and Participation in Placebo Controlled Randomized Clinical Trials (RCTs)
Description: Number of participants reporting attitudes and practices related to participation in placebo controlled RCTs during a semi-structured interview. Participants were selected for an interview based on their overall adherence rates, including those with excellent adherence throughout the study and those with lower adherence rates early or late in their participation. A trained female staff member conducted each 30-minute interview using an interview guide. Participants were asked about their attitudes toward participation in the study and research in general as HIV-infected women taking ART and at risk of preterm birth, but they were not specifically asked about their underlying knowledge of these conditions. Interviews were audio-taped, transcribed, and translated into English as necessary.
Time Frame: Late in pregnancy or postpartum
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Vaginal Progesterone | Placebo
Number analyzed (Participants) | 19 | 11
Participants
  Belief that being in the study prevented PTB | 15 | 6
  Belief that women might refuse a placebo RCT | 9 | 3
  Disclosed study participation to others | 19 | 10

5. Secondary Outcome: Acceptability of a Vaginal Medication to Prevent Preterm Birth
Description: Number of participants reporting specific attitudes about medications for the prevention of preterm birth (PTB), including acceptability of daily vaginal administration as measured on the Exit Satisfaction Survey using a Likert scale of five possible options ranging from strongly agree to strongly disagree. The form included a range of facial illustrations to facilitate comprehension of the answer choices, particularly for illiterate participants.
Time Frame: Visit 9.0 (36 weeks of gestation)
Population: 131 randomized participants who completed an exit satisfaction survey
Measure: Count of Participants; unit: Participants
Arm/Group | Vaginal Progesterone | Placebo
Number analyzed (Participants) | 67 | 64
Participants
  Happy that I took part in the study: Strongly disagree | 0 | 0
  Happy that I took part in the study: Disagree | 0 | 0
  Happy that I took part in the study: Neutral | 0 | 1
  Happy that I took part in the study: Agree | 1 | 3
  Happy that I took part in the study: Strongly agree | 66 | 60
  Did not mind taking daily vaginal medication: Strongly disagree | 0 | 0
  Did not mind taking daily vaginal medication: Disagree | 0 | 0
  Did not mind taking daily vaginal medication: Neutral | 0 | 1
  Did not mind taking daily vaginal medication: Agree | 9 | 3
  Did not mind taking daily vaginal medication: Strongly agree | 58 | 60
  Would choose daily vag med over wkly injection: Strongly disagree | 13 | 15
  Would choose daily vag med over wkly injection: Disagree | 3 | 0
  Would choose daily vag med over wkly injection: Neutral | 1 | 2
  Would choose daily vag med over wkly injection: Agree | 7 | 5
  Would choose daily vag med over wkly injection: Strongly agree | 43 | 42
  Other women would like to take med to stop PTB: Strongly disagree | 1 | 0
  Other women would like to take med to stop PTB: Disagree | 1 | 2
  Other women would like to take med to stop PTB: Neutral | 9 | 3
  Other women would like to take med to stop PTB: Agree | 16 | 15
  Other women would like to take med to stop PTB: Strongly agree | 40 | 44

6. Secondary Outcome: Reported Barriers to Adherence to Study Product
Description: Number of participants reporting challenges with taking the study medication as measured on the Exit Satisfaction Survey. The survey was administered by a study nurse who asked each participant what was the hardest part about taking the medication and presented all possible answer choices. Participant were asked to select only one answer.
Time Frame: Visit 9.0 (36 weeks of gestation)
Population: 131 randomized participants who completed an exit satisfaction survey
Measure: Count of Participants; unit: Participants
Arm/Group | Vaginal Progesterone | Placebo
Number analyzed (Participants) | 67 | 64
Participants
  Remembering to take it | 0 | 2
  Didn't like using the product | 0 | 0
  Obtaining refills at clinic | 0 | 0
  Disclosing participation to partner or family | 0 | 0
  Inserting the medication | 1 | 0
  Nothing was hard about taking the medication | 66 | 62

7. Secondary Outcome: Sensitivity, Specificity, and Predictive Value of Dose Diaries
Description: Comparison of self-reported adherence rates (Dose Diary/DD) and use of returned applicators measured by dye stain assay (DSA)
Time Frame: Enrollment through 36th gestational week, an overall total of up to 17 weeks
Population: Dose diaries completed by randomized participants returned at each follow-up visit, reported among participants who returned for at least 1 visit. Outcome assessed the reliability of dose diaries against DSA gold standard regardless of study arm to measure feasibility for future use. Estimates are presented in aggregate per original analysis plan.
Measure: Number (95% Confidence Interval); unit: Proportion of ppts correctly identified
Units Other Than Participants: Daily dose diaries
Groups:
- Daily Dose Diaries: Dose diaries completed by randomized participants returned at each follow-up visit
Arm/Group | Daily Dose Diaries
Number analyzed (Participants) | 137
Number analyzed (Daily dose diaries) | 12256
Proportion of ppts correctly identified
  Sensitivity Pr(DD+/DSA+) | 0.999 [0.999 to 1]
  Specificity Pr(DD-/DSA-) | 0.571 [0.521 to 0.619]
  Positive Predictive Value Pr(DSA+/DD+) | 0.985 [0.983 to 0.987]
  Negative Predictive Value Pr(DSA-/DD-) | 0.975 [0.946 to 0.991]

8. Secondary Outcome: Enrollment of Eligible Participants
Description: Number of eligible participants who enrolled in the study
Time Frame: Screening through Enrollment
Population: Women with a completed ultrasound who were eligible for study screening procedures
Measure: Count of Participants; unit: Participants
Groups:
- Women Eligible for Screening: Women eligible for study screening
Arm/Group | Women Eligible for Screening
Number analyzed (Participants) | 208
Participants
  Successfully Screened | 154
  Randomized | 140

9. Secondary Outcome: Ascertainment of Date of Delivery and Infant Vital Status
Description: Number of women for whom date of delivery and infant vital status at birth was ascertained
Time Frame: Visit 10.0 (Delivery)
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Vaginal Progesterone | Placebo
Number analyzed (Participants) | 70 | 70
Participants | 67 | 67

10. Secondary Outcome: Preliminary Efficacy
Description: Number of participants delivering before 34 and 37 completed weeks of gestation, grouped based on whether the participant went into labor spontaneously or was induced by a provider
Time Frame: Visit 10.0 (Delivery)
Measure: Count of Participants; unit: Participants
Arm/Group | Vaginal Progesterone | Placebo
Number analyzed (Participants) | 67 | 67
Participants
  Preterm birth <37 weeks | 9 | 10
  Spontaneous preterm birth <37 weeks | 8 | 10
  Preterm birth <34 weeks | 5 | 6
  Spontaneous preterm birth <34 weeks | 4 | 6

11. Secondary Outcome: Birth Weight
Description: Number of participants with neonates weighing less than 2500 grams at birth
Time Frame: Visit 10.0 (Delivery)
Population: Randomized participants with birth weight data ascertained
Measure: Count of Participants; unit: Participants
Arm/Group | Vaginal Progesterone | Placebo
Number analyzed (Participants) | 64 | 64
Participants | 9 | 12

12. Secondary Outcome: Stillbirth
Description: Number of participants who experienced a stillbirth
Time Frame: Visit 10.0 (Delivery)
Measure: Count of Participants; unit: Participants
Arm/Group | Vaginal Progesterone | Placebo
Number analyzed (Participants) | 67 | 67
Participants | 2 | 2

13. Secondary Outcome: Adverse Events
Description: Number of women experiencing a serious adverse event or event that resulted in study product discontinuation
Time Frame: Enrollment through Visit 10.0 (Delivery)
Measure: Count of Participants; unit: Participants
Arm/Group | Vaginal Progesterone | Placebo
Number analyzed (Participants) | 70 | 70
Participants
  Pre-eclampsia | 1 | 0
  Stillbirth | 2 | 2

ADVERSE EVENTS:
Time Frame: From the time of enrollment through delivery, a total of approximately 16-20 weeks.
Arm/Group | Vaginal Progesterone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/70
Serious Adverse Events (participants affected / at risk) | 3/70 | 2/70
Other Adverse Events (participants affected / at risk) | 34/70 | 29/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaginal Progesterone (N=70) | Placebo (N=70)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 2 (2)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaginal Progesterone (N=70) | Placebo (N=70)
Headache (General disorders) | 15 (15) | 10 (10)
Nausea/Vomiting (Gastrointestinal disorders) | 6 (6) | 6 (6)
Lower Abdominal Pain (General disorders) | 8 (8) | 5 (5)
Vaginal Itching/Burning (Reproductive system and breast disorders) | 5 (5) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/52/NCT02970552/Prot_SAP_000.pdf